CLINICAL TRIAL: NCT01294774
Title: A Multi-center, Double-blind, Placebo-controlled, Proof-of-concept Study to Evaluate the Efficacy and Tolerability of KRP203 in Patients With Active Subacute Cutaneous Lupus Erythematosus
Brief Title: Safety and Efficacy of KRP203 in Subacute Cutaneous Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CKRP203A2202; 2010-019689-10 (EudraCT Number)
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Subacute Cutaneous Lupus Erythematosus
Keywords: Lupus erythematosus; skin lupus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous | interventions — KRP-203

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- KRP203 - 1.2 mg (Experimental)
  Interventions: Drug: KRP203 - 1.2mg
- Placebo to KRP203 - 1.2 mg (Placebo Comparator)
  Interventions: Drug: Placebo to KRP203 - 1.2 mg

INTERVENTIONS:
Drug: KRP203 - 1.2mg
  Arms: KRP203 - 1.2 mg
Drug: Placebo to KRP203 - 1.2 mg
  Arms: Placebo to KRP203 - 1.2 mg

SUMMARY:
This study will assess the safety and efficacy of KRP203 in clinically active subacute cutaneous lupus erythematosus patients, who have demonstrated inadequate response to standard treatment, such as antimalarials.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients,18 to 65 years of age inclusive, who have been defined as having SCLE based on the typical clinical picture and the characteristic histopathological features as described by Sontheimer et al. at least three months before study entry (screening)

Exclusion Criteria:

1. Patients with preexisting nephritis, central nervous or pulmonary involvement or any major internal organ damage, either related or unrelated to lupus, which are deemed by the Investigator to be clinically significant. Patients having signs or symptoms of other autoimmune diseases such as systemic lupus erythematosus or Sjogren's syndrome are allowed to enter the study at the Investigator's discretion.
2. Patients who have been treated with:

   * immunoglobulins and/or monoclonal antibodies within 6 months prior to randomization.
   * rituximab, cyclophosphamide, or other immunosuppressive treatments with effects potentially lasting over 6 months, within 12 months prior to randomization.
   * a medium or high dose (≥ 1 mg prednisone or equivalent per body weight kg) corticosteroid therapy in the last 8 weeks prior to randomization.
   * antimalarial agents (hydroxychloroquine, chloroquine or quinacrine) in the last 6 weeks prior to randomization.
   * biologic therapies, such as etanercept, within the last 4 weeks prior to randomization.
   * any other immunosuppressive or immunomodulatory therapy such as methotrexate, azathioprine, cyclosporin A or mycophenolate, thalidomide, retinoids or dapsone in the last 4 weeks prior to randomization.
   * total lymphoid irradiation or bone marrow transplantation.
3. Pregnant, planning to get pregnant, and/or lactating females or males planning to father a child within time period of the study or subsequent exclusionary period.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of KRP203 in reduction of severity of symptoms, as measured using the activity score of the Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) | 12 weeks

SECONDARY OUTCOMES:
Safety and tolerability of oral KRP203 in patients with subacute cutaneous lupus erythematosus | 12 weeks
Steady-state blood concentrations of KRP203 and KRP203-Phosphate (KRP203-P) in SCLE patients | 12 weeks
Changes in the activity of SCLE using visual analogue scales for global skin health as assessed by the physician and the patient | 12 weeks
Measure the systemic features of SCLE using the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Germany (4):
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Tübingen
- Greece (2):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
- Italy (2):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Siena, SI